CLINICAL TRIAL: NCT04056767
Title: Measurement of Changes in the Digital Phenotype During Prolonged Exposure Therapy for PTSD Using Smart Watch
Brief Title: Changes in Digital Phenotype During PE Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nadav Goldental (Other)
Responsible Party: Sponsor-Investigator, Nadav Goldental, Principal investigator, The Chaim Sheba Medical Center
Organization: The Chaim Sheba Medical Center (Other)
Other Study IDs: 6269-19-SMC
Record Dates: First submitted 2019-08-06; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Imaginal PE
- Writing PE

SUMMARY:
PTSD is characterized by physiological changes, some of which are thought to be chronic, while others are observed in response to stressogenic stimuli. Prolonged Exposure (PE) therapy is a widely used protocol considered highly affective among individuals diagnosed with PTSD.

The current study is a non-interventional observational study, aimed at measuring changes in the digital phenotype of participants with PTSD during and following PE therapy. Physiological data will be collected using wearable sensors during the sessions, and participants will be assessed using questionnaires and psychiatric assessments before and after the completion of their imaginal or writing based PE therapy (10-15 sessions).

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis
* Proper ability to give informed consent

Exclusion Criteria:

* Active psychotic or suicidal symptoms
* Severe dissociative symptoms
* A traumatic brain injury (TBI) diagnosis
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (aged 18 and over) participants diagnosed with PTSD and undergoing PE therapy; 50 using imaginal PE and 50 using writing PE.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Heart Rate | 3 months
  Heart Rate and HRV (Heart Rate Variability)
Changes in Saturation | 3 months
  Changes in saturation SPO2 (oxygen saturation by pulse oximetry)
Changes in blood pressure | 3 months
  Changes in Continuous Blood Pressure
Changes in Pulse Pressure | 3 months
  Changes in Pulse Pressure
Changes in Respiratory rate | 3 months
  Changes in Respiratory rate
Changes in Stroke Volume | 3 months
  Changes in Stroke Volume
Changes in Systemic Vascular Resistance | 3 months
  Changes in Systemic Vascular Resistance
Changes in sweat | 3 months
  Changes in Sweat
Changes in Body Temperature | 3 months
  Changes in Body Temperature
Changes in Cardiac Output | 3 months
  Changes in Cardiac Output

SECONDARY OUTCOMES:
Correlation between changes in digital phenotype (multiple measures) | 3 months
  Correlation between changes in digital phenotype during the sessions and the clinical improvement according to the psychiatric evaluation and questionnaires.